CLINICAL TRIAL: NCT02230839
Title: Muscle Insulin Resistance In Aging
Brief Title: Muscle Insulin Resistance in Aging (Mirage)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth Translational Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: TRIMDFH 500423; NCT01808924 (obsolete NCT alias)
Record Dates: First submitted 2014-08-07; First posted 2014-09-03 (Estimated); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Insulin Resistance; Sarcopenia
Keywords: insulin resistance; muscle; health education; exercise
MeSH Terms: conditions — Insulin Resistance; Sarcopenia; Health Education; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise training protocol (Experimental)
  Interventions: Behavioral: Exercise
- Energy restriction-induced weight loss (Experimental)
  Interventions: Behavioral: Energy Restriction-Induced Weight Loss
- Health Education (No Intervention)

INTERVENTIONS:
Behavioral: Exercise — Participants will complete a progressive 6-month exercise training program, 4-5 days per week, 45 min per session (180 min per week), consisting mostly of walking (both outside and on an indoor treadmill) but with the option to include stationary cycling, elliptical and rowing machines, similar to what we have utilized previously to elicit significant improvements in insulin sensitivity in both middle-age and older adults (52-55). Beginning at week 8, these subjects will also perform 2 non-consecutive resistance exercise sessions per week, 30 min per session, focused on major muscle groups using resistance machines (total days of exercise will still be 4 to 5).
  Arms: Exercise training protocol
Behavioral: Energy Restriction-Induced Weight Loss — The goal of the weight loss intervention will be to produce a weight loss of 10% body weight. A reduction of 500-1000 kcal/day - based on baseline weight -and low fat (<30% of calories from fat) diet will be used as part of the weight loss intervention.
  Arms: Energy restriction-induced weight loss

SUMMARY:
The purpose of this study is to provide information regarding potential factors underlying metabolic dysfunction, insulin resistance, and loss of muscle mass in aging muscle.

DETAILED DESCRIPTION:
Study Objectives:

1. To determine the effects of diet-induced weight loss with and without the addition of exercise on mitochondrial biogenesis and energetic capacity, cellular redox state and insulin resistance.
2. To determine the effects of diet-induced weight loss with and without the addition of exercise on intramyocellular lipid profiles.
3. To determine the effects of diet-induced weight loss with and without exercise on skeletal muscle proteins mediating a program of autophagy and either loss or maintenance of muscle mass.

ELIGIBILITY:
Inclusion Criteria:

* 65-80 years of age
* Stable weight (No Gain/Loss of >10 lbs in 6 months)
* Sedentary (≤ 1 continuous exercise/week)
* Non-smoker
* BMI ≥ 30 kg/m2
* Resting Blood Pressure ≤ 150 millimeters of mercury systolic and ≤ 95 millimeters of mercury diastolic
* Note from Primary care physician/Cardiologist for exercise clearance if positive stress test symptoms were observed from exercise test
* Must be willing to washout for 14 days from all diabetes medication and independent in self blood glucose monitoring during the washout periods (those with diabetes only)

Exclusion Criteria:

* Clinically significant cardiovascular disease including history of myocardial infarction, within the past year
* Peripheral Vascular Disease
* Hepatic, renal, muscular/neuromuscular, or active hematologic/oncologic disease
* Clinically diminished pulse
* Presence of bruits in lower extremities
* Previous history of pulmonary emboli
* Peripheral Neuropathy

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-06; Primary Completion 2023-12-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Measure of intramyocellular lipids | Visit 3 ~22 hours
  A percutaneous muscle biopsy of the vastus lateralis will be obtained, and the intramyocellular lipids will be measured by high-performance liquid chromatography-tandem mass spectrometry.

SECONDARY OUTCOMES:
Measure of insulin sensitivity | Visit 3 ~22 hours
  Insulin sensitivity will be measured using an intravenous catheter (glucose clamps) that will be placed in the antecubital vein for subsequent insulin and glucose infusions and for stable isotope infusions. This will measure insulin-stimulated changes in insulin signaling proteins and metabolism.

OTHER OUTCOMES:
Measure muscle strength and power | Visit 2 (baseline) and 6 months
  Muscle strength and power will be measured in participants who have successfully completed all screening procedures.
  Measurement is obtained using a short physical performance battery, knee extension, and muscle power testing using a pneumatic-driven dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Bret Goodpaster, PhD, Principal Investigator — Translational Research Institute for Metabolism and Diabetes
Locations (1):
- Translational Research Institute for Metabolism and Diabetes, Orlando, Florida, United States

REFERENCES:
- [Background] Evans W. Functional and metabolic consequences of sarcopenia. J Nutr. 1997 May;127(5 Suppl):998S-1003S. doi: 10.1093/jn/127.5.998S. PMID 9164283
- [Background] Evans WJ, Campbell WW. Sarcopenia and age-related changes in body composition and functional capacity. J Nutr. 1993 Feb;123(2 Suppl):465-8. doi: 10.1093/jn/123.suppl_2.465. PMID 8429405
- [Background] Rosenberg IH. Sarcopenia: origins and clinical relevance. J Nutr. 1997 May;127(5 Suppl):990S-991S. doi: 10.1093/jn/127.5.990S. PMID 9164280
- [Background] Ogden CL, Carroll MD, Curtin LR, McDowell MA, Tabak CJ, Flegal KM. Prevalence of overweight and obesity in the United States, 1999-2004. JAMA. 2006 Apr 5;295(13):1549-55. doi: 10.1001/jama.295.13.1549. PMID 16595758
- [Background] Villareal DT, Apovian CM, Kushner RF, Klein S; American Society for Nutrition; NAASO, The Obesity Society. Obesity in older adults: technical review and position statement of the American Society for Nutrition and NAASO, The Obesity Society. Am J Clin Nutr. 2005 Nov;82(5):923-34. doi: 10.1093/ajcn/82.5.923. PMID 16280421
- [Background] Goodpaster BH, Carlson CL, Visser M, Kelley DE, Scherzinger A, Harris TB, Stamm E, Newman AB. Attenuation of skeletal muscle and strength in the elderly: The Health ABC Study. J Appl Physiol (1985). 2001 Jun;90(6):2157-65. doi: 10.1152/jappl.2001.90.6.2157. PMID 11356778
- [Background] Park SW, Goodpaster BH, Lee JS, Kuller LH, Boudreau R, de Rekeneire N, Harris TB, Kritchevsky S, Tylavsky FA, Nevitt M, Cho YW, Newman AB; Health, Aging, and Body Composition Study. Excessive loss of skeletal muscle mass in older adults with type 2 diabetes. Diabetes Care. 2009 Nov;32(11):1993-7. doi: 10.2337/dc09-0264. Epub 2009 Jun 23. PMID 19549734
- [Background] Petersen KF, Befroy D, Dufour S, Dziura J, Ariyan C, Rothman DL, DiPietro L, Cline GW, Shulman GI. Mitochondrial dysfunction in the elderly: possible role in insulin resistance. Science. 2003 May 16;300(5622):1140-2. doi: 10.1126/science.1082889. PMID 12750520
- [Background] Amati F, Dube JJ, Coen PM, Stefanovic-Racic M, Toledo FG, Goodpaster BH. Physical inactivity and obesity underlie the insulin resistance of aging. Diabetes Care. 2009 Aug;32(8):1547-9. doi: 10.2337/dc09-0267. Epub 2009 Apr 28. PMID 19401446
- [Background] Kelley DE, Goodpaster B, Wing RR, Simoneau JA. Skeletal muscle fatty acid metabolism in association with insulin resistance, obesity, and weight loss. Am J Physiol. 1999 Dec;277(6):E1130-41. doi: 10.1152/ajpendo.1999.277.6.E1130. PMID 10600804
- [Background] Kelley DE, Mintun MA, Watkins SC, Simoneau JA, Jadali F, Fredrickson A, Beattie J, Theriault R. The effect of non-insulin-dependent diabetes mellitus and obesity on glucose transport and phosphorylation in skeletal muscle. J Clin Invest. 1996 Jun 15;97(12):2705-13. doi: 10.1172/JCI118724. PMID 8675680
- [Background] Lillioja S, Bogardus C. Obesity and insulin resistance: lessons learned from the Pima Indians. Diabetes Metab Rev. 1988 Aug;4(5):517-40. doi: 10.1002/dmr.5610040508. PMID 3061759
- [Background] Devlin JT. Effects of exercise on insulin sensitivity in humans. Diabetes Care. 1992 Nov;15(11):1690-3. doi: 10.2337/diacare.15.11.1690. PMID 1468302
- [Background] Bogardus C. Insulin resistance in the pathogenesis of NIDDM in Pima Indians. Diabetes Care. 1993 Jan;16(1):228-31. doi: 10.2337/diacare.16.1.228. PMID 8422780
- [Background] Haffner SM, Valdez RA, Hazuda HP, Mitchell BD, Morales PA, Stern MP. Prospective analysis of the insulin-resistance syndrome (syndrome X). Diabetes. 1992 Jun;41(6):715-22. doi: 10.2337/diab.41.6.715. PMID 1587398
- [Background] Rizza RA, Mandarino LJ, Gerich JE. Mechanism and significance of insulin resistance in non-insulin-dependent diabetes mellitus. Diabetes. 1981 Dec;30(12):990-5. doi: 10.2337/diab.30.12.990. PMID 7030834
- [Background] Chavez JA, Knotts TA, Wang LP, Li G, Dobrowsky RT, Florant GL, Summers SA. A role for ceramide, but not diacylglycerol, in the antagonism of insulin signal transduction by saturated fatty acids. J Biol Chem. 2003 Mar 21;278(12):10297-303. doi: 10.1074/jbc.M212307200. Epub 2003 Jan 13. PMID 12525490
- [Background] Stratford S, Hoehn KL, Liu F, Summers SA. Regulation of insulin action by ceramide: dual mechanisms linking ceramide accumulation to the inhibition of Akt/protein kinase B. J Biol Chem. 2004 Aug 27;279(35):36608-15. doi: 10.1074/jbc.M406499200. Epub 2004 Jun 25. PMID 15220355
- [Background] Turinsky J, O'Sullivan DM, Bayly BP. 1,2-Diacylglycerol and ceramide levels in insulin-resistant tissues of the rat in vivo. J Biol Chem. 1990 Oct 5;265(28):16880-5. PMID 2211599
- [Background] Holland WL, Brozinick JT, Wang LP, Hawkins ED, Sargent KM, Liu Y, Narra K, Hoehn KL, Knotts TA, Siesky A, Nelson DH, Karathanasis SK, Fontenot GK, Birnbaum MJ, Summers SA. Inhibition of ceramide synthesis ameliorates glucocorticoid-, saturated-fat-, and obesity-induced insulin resistance. Cell Metab. 2007 Mar;5(3):167-79. doi: 10.1016/j.cmet.2007.01.002. PMID 17339025
- [Background] Adams JM 2nd, Pratipanawatr T, Berria R, Wang E, DeFronzo RA, Sullards MC, Mandarino LJ. Ceramide content is increased in skeletal muscle from obese insulin-resistant humans. Diabetes. 2004 Jan;53(1):25-31. doi: 10.2337/diabetes.53.1.25. PMID 14693694
- [Background] Itani SI, Ruderman NB, Schmieder F, Boden G. Lipid-induced insulin resistance in human muscle is associated with changes in diacylglycerol, protein kinase C, and IkappaB-alpha. Diabetes. 2002 Jul;51(7):2005-11. doi: 10.2337/diabetes.51.7.2005. PMID 12086926
- [Background] Bruce CR, Thrush AB, Mertz VA, Bezaire V, Chabowski A, Heigenhauser GJ, Dyck DJ. Endurance training in obese humans improves glucose tolerance and mitochondrial fatty acid oxidation and alters muscle lipid content. Am J Physiol Endocrinol Metab. 2006 Jul;291(1):E99-E107. doi: 10.1152/ajpendo.00587.2005. Epub 2006 Feb 7. PMID 16464906
- [Background] Bergman BC, Perreault L, Hunerdosse DM, Koehler MC, Samek AM, Eckel RH. Increased intramuscular lipid synthesis and low saturation relate to insulin sensitivity in endurance-trained athletes. J Appl Physiol (1985). 2010 May;108(5):1134-41. doi: 10.1152/japplphysiol.00684.2009. Epub 2010 Mar 18. PMID 20299618
- [Background] Perreault L, Bergman BC, Hunerdosse DM, Playdon MC, Eckel RH. Inflexibility in intramuscular triglyceride fractional synthesis distinguishes prediabetes from obesity in humans. Obesity (Silver Spring). 2010 Aug;18(8):1524-31. doi: 10.1038/oby.2009.454. Epub 2009 Dec 24. PMID 20035285
- [Background] Bergman BC, Perreault L, Hunerdosse DM, Koehler MC, Samek AM, Eckel RH. Intramuscular lipid metabolism in the insulin resistance of smoking. Diabetes. 2009 Oct;58(10):2220-7. doi: 10.2337/db09-0481. Epub 2009 Jul 6. PMID 19581421
- [Background] Lowell BB, Shulman GI. Mitochondrial dysfunction and type 2 diabetes. Science. 2005 Jan 21;307(5708):384-7. doi: 10.1126/science.1104343. PMID 15662004
- [Background] Holloszy JO. "Deficiency" of mitochondria in muscle does not cause insulin resistance. Diabetes. 2013 Apr;62(4):1036-40. doi: 10.2337/db12-1107. PMID 23520283
- [Background] Li J, Romestaing C, Han X, Li Y, Hao X, Wu Y, Sun C, Liu X, Jefferson LS, Xiong J, Lanoue KF, Chang Z, Lynch CJ, Wang H, Shi Y. Cardiolipin remodeling by ALCAT1 links oxidative stress and mitochondrial dysfunction to obesity. Cell Metab. 2010 Aug 4;12(2):154-65. doi: 10.1016/j.cmet.2010.07.003. PMID 20674860
- [Background] Lee HY, Choi CS, Birkenfeld AL, Alves TC, Jornayvaz FR, Jurczak MJ, Zhang D, Woo DK, Shadel GS, Ladiges W, Rabinovitch PS, Santos JH, Petersen KF, Samuel VT, Shulman GI. Targeted expression of catalase to mitochondria prevents age-associated reductions in mitochondrial function and insulin resistance. Cell Metab. 2010 Dec 1;12(6):668-74. doi: 10.1016/j.cmet.2010.11.004. PMID 21109199
- [Background] Reznick RM, Zong H, Li J, Morino K, Moore IK, Yu HJ, Liu ZX, Dong J, Mustard KJ, Hawley SA, Befroy D, Pypaert M, Hardie DG, Young LH, Shulman GI. Aging-associated reductions in AMP-activated protein kinase activity and mitochondrial biogenesis. Cell Metab. 2007 Feb;5(2):151-6. doi: 10.1016/j.cmet.2007.01.008. PMID 17276357
- [Background] Masiero E, Agatea L, Mammucari C, Blaauw B, Loro E, Komatsu M, Metzger D, Reggiani C, Schiaffino S, Sandri M. Autophagy is required to maintain muscle mass. Cell Metab. 2009 Dec;10(6):507-15. doi: 10.1016/j.cmet.2009.10.008. PMID 19945408
- [Background] Wenz T, Rossi SG, Rotundo RL, Spiegelman BM, Moraes CT. Increased muscle PGC-1alpha expression protects from sarcopenia and metabolic disease during aging. Proc Natl Acad Sci U S A. 2009 Dec 1;106(48):20405-10. doi: 10.1073/pnas.0911570106. Epub 2009 Nov 16. PMID 19918075 (Retraction: PMID 27994157 Proc Natl Acad Sci U S A. 2016 Dec 19;:)
- [Background] Romanello V, Guadagnin E, Gomes L, Roder I, Sandri C, Petersen Y, Milan G, Masiero E, Del Piccolo P, Foretz M, Scorrano L, Rudolf R, Sandri M. Mitochondrial fission and remodelling contributes to muscle atrophy. EMBO J. 2010 May 19;29(10):1774-85. doi: 10.1038/emboj.2010.60. Epub 2010 Apr 16. PMID 20400940
- [Background] Civitarese AE, Carling S, Heilbronn LK, Hulver MH, Ukropcova B, Deutsch WA, Smith SR, Ravussin E; CALERIE Pennington Team. Calorie restriction increases muscle mitochondrial biogenesis in healthy humans. PLoS Med. 2007 Mar;4(3):e76. doi: 10.1371/journal.pmed.0040076. PMID 17341128
- [Background] Fontana L, Villareal DT, Weiss EP, Racette SB, Steger-May K, Klein S, Holloszy JO; Washington University School of Medicine CALERIE Group. Calorie restriction or exercise: effects on coronary heart disease risk factors. A randomized, controlled trial. Am J Physiol Endocrinol Metab. 2007 Jul;293(1):E197-202. doi: 10.1152/ajpendo.00102.2007. Epub 2007 Mar 27. PMID 17389710
- [Background] Heilbronn LK, de Jonge L, Frisard MI, DeLany JP, Larson-Meyer DE, Rood J, Nguyen T, Martin CK, Volaufova J, Most MM, Greenway FL, Smith SR, Deutsch WA, Williamson DA, Ravussin E; Pennington CALERIE Team. Effect of 6-month calorie restriction on biomarkers of longevity, metabolic adaptation, and oxidative stress in overweight individuals: a randomized controlled trial. JAMA. 2006 Apr 5;295(13):1539-48. doi: 10.1001/jama.295.13.1539. PMID 16595757
- [Background] Santanasto AJ, Glynn NW, Newman MA, Taylor CA, Brooks MM, Goodpaster BH, Newman AB. Impact of weight loss on physical function with changes in strength, muscle mass, and muscle fat infiltration in overweight to moderately obese older adults: a randomized clinical trial. J Obes. 2011;2011:516576. doi: 10.1155/2011/516576. Epub 2010 Oct 10. PMID 20953373
- [Background] Messier SP, Loeser RF, Mitchell MN, Valle G, Morgan TP, Rejeski WJ, Ettinger WH. Exercise and weight loss in obese older adults with knee osteoarthritis: a preliminary study. J Am Geriatr Soc. 2000 Sep;48(9):1062-72. doi: 10.1111/j.1532-5415.2000.tb04781.x. PMID 10983905
- [Background] Weiss EP, Racette SB, Villareal DT, Fontana L, Steger-May K, Schechtman KB, Klein S, Ehsani AA, Holloszy JO; Washington University School of Medicine CALERIE Group. Lower extremity muscle size and strength and aerobic capacity decrease with caloric restriction but not with exercise-induced weight loss. J Appl Physiol (1985). 2007 Feb;102(2):634-40. doi: 10.1152/japplphysiol.00853.2006. Epub 2006 Nov 9. PMID 17095635
- [Background] Goodpaster BH, He J, Watkins S, Kelley DE. Skeletal muscle lipid content and insulin resistance: evidence for a paradox in endurance-trained athletes. J Clin Endocrinol Metab. 2001 Dec;86(12):5755-61. doi: 10.1210/jcem.86.12.8075. PMID 11739435
- [Background] Kelley DE, He J, Menshikova EV, Ritov VB. Dysfunction of mitochondria in human skeletal muscle in type 2 diabetes. Diabetes. 2002 Oct;51(10):2944-50. doi: 10.2337/diabetes.51.10.2944. PMID 12351431
- [Background] Ritov VB, Menshikova EV, Kelley DE. Analysis of cardiolipin in human muscle biopsy. J Chromatogr B Analyt Technol Biomed Life Sci. 2006 Feb 2;831(1-2):63-71. doi: 10.1016/j.jchromb.2005.11.031. Epub 2005 Dec 6. PMID 16337440
- [Background] Ritov VB, Menshikova EV, Kelley DE. High-performance liquid chromatography-based methods of enzymatic analysis: electron transport chain activity in mitochondria from human skeletal muscle. Anal Biochem. 2004 Oct 1;333(1):27-38. doi: 10.1016/j.ab.2004.05.014. PMID 15351277
- [Background] Dube JJ, Amati F, Stefanovic-Racic M, Toledo FG, Sauers SE, Goodpaster BH. Exercise-induced alterations in intramyocellular lipids and insulin resistance: the athlete's paradox revisited. Am J Physiol Endocrinol Metab. 2008 May;294(5):E882-8. doi: 10.1152/ajpendo.00769.2007. Epub 2008 Mar 4. PMID 18319352
- [Background] Goodpaster BH, Katsiaras A, Kelley DE. Enhanced fat oxidation through physical activity is associated with improvements in insulin sensitivity in obesity. Diabetes. 2003 Sep;52(9):2191-7. doi: 10.2337/diabetes.52.9.2191. PMID 12941756
- [Background] Pruchnic R, Katsiaras A, He J, Kelley DE, Winters C, Goodpaster BH. Exercise training increases intramyocellular lipid and oxidative capacity in older adults. Am J Physiol Endocrinol Metab. 2004 Nov;287(5):E857-62. doi: 10.1152/ajpendo.00459.2003. Epub 2004 Jun 29. PMID 15226098
- [Background] Dube JJ, Amati F, Toledo FG, Stefanovic-Racic M, Rossi A, Coen P, Goodpaster BH. Effects of weight loss and exercise on insulin resistance, and intramyocellular triacylglycerol, diacylglycerol and ceramide. Diabetologia. 2011 May;54(5):1147-56. doi: 10.1007/s00125-011-2065-0. Epub 2011 Feb 17. PMID 21327867
- [Background] Goodpaster BH, Chomentowski P, Ward BK, Rossi A, Glynn NW, Delmonico MJ, Kritchevsky SB, Pahor M, Newman AB. Effects of physical activity on strength and skeletal muscle fat infiltration in older adults: a randomized controlled trial. J Appl Physiol (1985). 2008 Nov;105(5):1498-503. doi: 10.1152/japplphysiol.90425.2008. Epub 2008 Sep 25. PMID 18818386
- [Background] LIFE Study Investigators; Pahor M, Blair SN, Espeland M, Fielding R, Gill TM, Guralnik JM, Hadley EC, King AC, Kritchevsky SB, Maraldi C, Miller ME, Newman AB, Rejeski WJ, Romashkan S, Studenski S. Effects of a physical activity intervention on measures of physical performance: Results of the lifestyle interventions and independence for Elders Pilot (LIFE-P) study. J Gerontol A Biol Sci Med Sci. 2006 Nov;61(11):1157-65. doi: 10.1093/gerona/61.11.1157. PMID 17167156
- [Background] Goodpaster BH, Theriault R, Watkins SC, Kelley DE. Intramuscular lipid content is increased in obesity and decreased by weight loss. Metabolism. 2000 Apr;49(4):467-72. doi: 10.1016/s0026-0495(00)80010-4. PMID 10778870
- [Background] Gnaiger E. Capacity of oxidative phosphorylation in human skeletal muscle: new perspectives of mitochondrial physiology. Int J Biochem Cell Biol. 2009 Oct;41(10):1837-45. doi: 10.1016/j.biocel.2009.03.013. Epub 2009 Apr 2. PMID 19467914
- [Background] Hutter E, Unterluggauer H, Garedew A, Jansen-Durr P, Gnaiger E. High-resolution respirometry--a modern tool in aging research. Exp Gerontol. 2006 Jan;41(1):103-9. doi: 10.1016/j.exger.2005.09.011. Epub 2005 Nov 23. PMID 16309877
- [Background] Goodpaster BH, Kelley DE, Wing RR, Meier A, Thaete FL. Effects of weight loss on regional fat distribution and insulin sensitivity in obesity. Diabetes. 1999 Apr;48(4):839-47. doi: 10.2337/diabetes.48.4.839. PMID 10102702
- [Background] Goodpaster BH, Thaete FL, Kelley DE. Thigh adipose tissue distribution is associated with insulin resistance in obesity and in type 2 diabetes mellitus. Am J Clin Nutr. 2000 Apr;71(4):885-92. doi: 10.1093/ajcn/71.4.885. PMID 10731493
- [Background] Toledo FG, Menshikova EV, Ritov VB, Azuma K, Radikova Z, DeLany J, Kelley DE. Effects of physical activity and weight loss on skeletal muscle mitochondria and relationship with glucose control in type 2 diabetes. Diabetes. 2007 Aug;56(8):2142-7. doi: 10.2337/db07-0141. Epub 2007 May 29. PMID 17536063
- [Background] Toledo FG, Watkins S, Kelley DE. Changes induced by physical activity and weight loss in the morphology of intermyofibrillar mitochondria in obese men and women. J Clin Endocrinol Metab. 2006 Aug;91(8):3224-7. doi: 10.1210/jc.2006-0002. Epub 2006 May 9. PMID 16684829
- [Background] Bielawski J, Szulc ZM, Hannun YA, Bielawska A. Simultaneous quantitative analysis of bioactive sphingolipids by high-performance liquid chromatography-tandem mass spectrometry. Methods. 2006 Jun;39(2):82-91. doi: 10.1016/j.ymeth.2006.05.004. PMID 16828308
- [Background] Sun D, Cree MG, Wolfe RR. Quantification of the concentration and 13C tracer enrichment of long-chain fatty acyl-coenzyme A in muscle by liquid chromatography/mass spectrometry. Anal Biochem. 2006 Feb 1;349(1):87-95. doi: 10.1016/j.ab.2005.10.006. Epub 2005 Oct 26. PMID 16307720
- [Background] Jubrias SA, Crowther GJ, Shankland EG, Gronka RK, Conley KE. Acidosis inhibits oxidative phosphorylation in contracting human skeletal muscle in vivo. J Physiol. 2003 Dec 1;553(Pt 2):589-99. doi: 10.1113/jphysiol.2003.045872. Epub 2003 Sep 26. PMID 14514869
- [Background] Blei ML, Conley KE, Kushmerick MJ. Separate measures of ATP utilization and recovery in human skeletal muscle. J Physiol. 1993 Jun;465:203-22. doi: 10.1113/jphysiol.1993.sp019673. PMID 8024651
- See also: Florida Hospital Translational Research Institute for Metabolism and Diabetes — http://www.tri-md.org